CLINICAL TRIAL: NCT07111403
Title: Remineralization Potential of Different Remineralizing Agents on Initial Enamel Caries: Laboratory Evaluations and Two-year Randomized Clinical Trial
Brief Title: Clinical Evaluation of Remineralizing Potential of Remineralizing Agents on WSLs Managment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0108024CD
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-09

CONDITIONS: Initial Dental Caries; White Spot Lesion of Tooth

STUDY DESIGN:
Intervention Model Description: Participants in each group received one remineralizing material according to manufacture's instructions or previous studies' recommendations after tooth isolation.
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAP fluoride plus (Active Comparator): Participants in this group received P11-4 (Curodont Repair™, Biomedical products for tooth preservation) only at baseline. First, the tooth was completely isolated using rubber dam followed by cleaning of the tooth surface with sodium hypochlorite 2% for 20 s, acid etching with phosphoric acid gel 35-37% for 20 s, rinsing and drying.
  Interventions: Procedure: SAP fluoride plus
- 10% n-HAp (Active Comparator): A Low-speed handpiece was used to clean the tooth surface with fluoride-free pumice (Pumice powder extra fine, SSWhite, Rio de Janeiro, Brazil) after tooth isolation, rinsing, and drying. after that the material was applied
  Interventions: Procedure: 10% n-HAp.
- 10% n-BAG. (Active Comparator): A Low-speed handpiece was used to clean the tooth surface with fluoride-free pumice (Pumice powder extra fine, SSWhite, Rio de Janeiro, Brazil) after tooth isolation, rinsing, and drying. after that the material was applied
  Interventions: Procedure: 10% n-BAG.
- Flour Protector S (Active Comparator): The teeth were dried and a very thin coat of the varnish was applied and allowed to dry for 20 s.
  Interventions: Procedure: Flour Protector S

INTERVENTIONS:
Procedure: SAP fluoride plus — The agent was applied by removing the safety clip, activating the applicator and squeezing out the sponge above the lesion and the solution was left to diffuse for 5 min.the patients were instructed to eat only soft foods and avoid hot liquids for two hours. Also, they were educated and motivated about the importance of oral hygiene.
  Arms: SAP fluoride plus
Procedure: 10% n-HAp. — the pastes were applied using micro brushes. The excess was removed after four minutes with a cotton swab. The subjects were advised not to drink or eat for 30 minutes after the treatment. The treatment was applied once every week for a period of four weeks.they instructed to adhere to oral hygiene measures.
  Arms: 10% n-HAp
Procedure: 10% n-BAG. — the pastes were applied using micro brushes. The excess was removed after four minutes with a cotton swab. The subjects were advised not to drink or eat for 30 minutes after the treatment. The treatment was applied once every week for a period of four weeks. patients instructed to adhere to oral hygiene measures.
  Arms: 10% n-BAG.
Procedure: Flour Protector S — After application of varnish, the patient was instructed to avoid abrasive diet for the rest of the day and not brush or floss until the next morning. The treatment was done at baseline and after 6 months.
  Arms: Flour Protector S

SUMMARY:
To evaluate and compare the clinical effect of four different remineralizing agents on initial enamel caries after a two years follow up.

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a double-blinded randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation. The trial will follow a parallel-arm design.A young- age patients , who are seeking dental treatment, will be enrolled in the study. The participants will be recruited from the Operative Department clinic at the Facultyof Dentistry, University of Mansoura. The study will focus on initial enamel caries on buccal or labial surfaces of permenant teeth.rior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The study is scheduled to be conducted from September 2024 to September 2026. The form and protocol of the study will be approved by Mansoura University's ethics committee before initiation.Sample size calculation was based on mean NYVAD scores between studied groups retrieved from previous research that most similar to our research using G power program version 3.1.9.7 to calculate sample size based on expected difference of 31% ,using 2-tailed test , α error =0.05 and power = 80.0% , the total calculated sample size will be at least 30 in each group with each patient having at least one active lesion.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have at least one visible initial enamel caries in the permanent teeth
* Only lesions with ICDAS II score of 1 or 2 could be included
* The patients must have good oral hygiene

Exclusion Criteria:

* patients receiving tetracyclines, any other medication known to stain teeth - Patients had fluoride application less than 3 months before the study
* Teeth which have microcavities or dentinal involvement due to loss of enamel - Teeth that have discoloration, enamel hypoplasia or fluorosis.

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
ICDAS II scores | assessment will be done at baseline and after 3, 6, 12 and 24 months.
  Remineralization will be assessed using visual tactile assessment of white spot lesions based on change in ICDAS II scores (reduction from score 2 to 1, or from score 1 to 0).

SECONDARY OUTCOMES:
DIAGNOdent score | assessment will be done at baseline and after 3, 6, 12 and 24 months.
  Remineralization will be assessed using The DIAGNOdent score which ranges from 0 to 99 with higher score indicating deeper caries. A decrease in value indicates regression of the carious lesion, whereas an increase indicates progression.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A Arisha, Ass Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt
Locations (1):
- Faculty of Dentistry, Mansoura University, Egypt, Al Mansurah, Egypt